CLINICAL TRIAL: NCT02308514
Title: Does Adding Cryostimulation to Conservative Care Help in Managing Chronic Lateral Epicondylitis? a Pilote Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Nadia Richer, Nadia Richer, M.Sc., DC, clinician professor, Université du Québec à Trois-Rivières
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CER-14-203-07.08
Record Dates: First submitted 2014-11-26; First posted 2014-12-04 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Lateral Epicondylitis
Keywords: cryostimulation
MeSH Terms: conditions — Tennis Elbow | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- conservative care (Active Comparator): this group of patients will receive the conservative care: myofascial point release and radial head mobilisation
  Interventions: Other: conservative care
- cryostimulation (Experimental): this group of patients will receive the conservative care :myofascial point release and radial haed mobilisation and the cryostimulation (30-40 second of cold air application (-70 celsius degree) in order to lower skin temperature around the lateral epicondyle at 4 celsius degree.
  Interventions: Device: cryostimulation; Other: conservative care

INTERVENTIONS:
Device: cryostimulation — pressurized cold air (-70 celsius degree) is blown on the skin surface surrounding the lateral epicondyle, creating a rapid decrease in ski temperature. In a 30-40 sec exposition, skin temperature can drop to 4 celsius degree. this rapid decrease is presumed to have a positive healing effect.
  Arms: cryostimulation
Other: conservative care — manual treatment of localized tender and painful myofascial areas in the muscles surrounding the forearm and mobilization of the radial head.
  Other Names: myofascial release

SUMMARY:
In this study the investigators want to measure the impact or effects of adding cryostimulation to the conservative care of chronic lateral epicondylitis. The rapid fall in skin temperature above the injured tissues is presume to have a positive effect in the healing process. The combination of conservative care and cryostimulation could then be appreciated. The investigators chose to measure these effects with 3 elements: visual analog pain scale, validated elbow questionnaire and pain free grip strength. This pilot study consist in a two arm design, each arm including 15 patients.

DETAILED DESCRIPTION:
Lateral epicondylitis is one of the most prevalent upper limb conditions that can affect up to 1-3% of the active population. Invalidity and health care costs incurred by this condition are posing a real challenge to our societies knowing that the natural history of the lateral epicondylitis can last from 1 to 2 years. Many therapies have been tested and so far none has proven conclusive when used alone so far (Blanchette and Normand 2011). The use of cryostimulation is widespread in the sport scene without strong literature supporting its evidence. The aim of this study is to quantify the effects of cryostimulation when added to conservative care in the treatment of chronic lateral epicondylitis.

Thirty (30) patients will be divided randomly in two groups:

* The control group (n=15) will receive conservative care including myofascial trigger points (involved forearm) and radial head mobilisations (Bergmann & Peterson, 2010).
* The experimental group (n=15) will receive the cryostimulation and the conservative treatment as mentioned above.

A total of eight treatments will be given to each patient; the whole protocol lasting four to six weeks. The treatments will be delivered by experienced and trained clinicians in cryostimulation and myofascial treatment protocols.

The effects of the two treatment protocols will be monitored by a validated elbow questionnaire (PRTEE, (Rompe, Overend et al. 2007)), a visual analog pain scale and the pain free grip strength at three moments: at inclusion, at the ninth visit and 3 months after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must have pain at lateral elbow (lateral epicondylitis) for at least six months
* Pain must not come from trauma
* Painful palpation of the lateral epicondyle
* At least one out of two positive test: Cozen's, Mill's

Exclusion Criteria:

* Fibromyalgia
* Diabetes
* Patient taking more than three medications at the time of inclusion
* Cervical radiculopathy
* Painful shoulder
* Cold intolerance / allergies
* Smoking
* Cortisone infiltration at the painful lateral epicondyle in the month previous to the inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Pain Scale | at inclusion - ninth visit - 3 months after last treatment
  Subjects will be asked to rate their average pain for the last 24 hours on a scale ranging from 0 to 10

SECONDARY OUTCOMES:
pain free grip strength | at inclusion - ninth visit - 3 months after last treatment
  we will use a hand-held dynamometer to mesure the painfree grip strength of the subjets. Subjects will be asked to gradually increase the grip stregth while the elbow is extented and arm along side of the body. They will be asked to stop when pain is felt. We will take three mesures with each elbow, left and right.

OTHER OUTCOMES:
Patient Rated Tennis Elbow | at inclusion - ninth visit - 3 months after last treatment
  The questionnaire will be filled in by patients at the beginning of the three evaluations: inclusion, ninth visit and 3 months after last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Richer Richer, M.Sc., Principal Investigator — Clinique universitaire de chiropratique
Locations (1):
- Clinique universitaire de chiropratique, Trois-Rivières, Quebec, Canada

REFERENCES:
- [Background] Blanchette MA, Normand MC. Impairment assessment of lateral epicondylitis through electromyography and dynamometry. J Can Chiropr Assoc. 2011 Jun;55(2):96-106. PMID 21629462
- [Background] Rompe JD, Overend TJ, MacDermid JC. Validation of the Patient-rated Tennis Elbow Evaluation Questionnaire. J Hand Ther. 2007 Jan-Mar;20(1):3-10; quiz 11. doi: 10.1197/j.jht.2006.10.003. PMID 17254903
- [Background] Mourot L, Cluzeau C, Regnard J. Hyperbaric gaseous cryotherapy: effects on skin temperature and systemic vasoconstriction. Arch Phys Med Rehabil. 2007 Oct;88(10):1339-43. doi: 10.1016/j.apmr.2007.06.771. PMID 17908579
- [Background] Dingemanse R, Randsdorp M, Koes BW, Huisstede BM. Evidence for the effectiveness of electrophysical modalities for treatment of medial and lateral epicondylitis: a systematic review. Br J Sports Med. 2014 Jun;48(12):957-65. doi: 10.1136/bjsports-2012-091513. Epub 2013 Jan 18. PMID 23335238
- [Background] Coombes BK, Bisset L, Vicenzino B. Thermal hyperalgesia distinguishes those with severe pain and disability in unilateral lateral epicondylalgia. Clin J Pain. 2012 Sep;28(7):595-601. doi: 10.1097/AJP.0b013e31823dd333. PMID 22699135